CLINICAL TRIAL: NCT00001621
Title: Evaluation and Treatment of Pulmonary Patients Not Participating in Research (Training Protocol)
Brief Title: Evaluation and Treatment of Patients With Lung Disease Not Participating in Research
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970061; 97-H-0061
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Disease
Keywords: Teaching; Pulmonary Disease; Routine Testing; Medically Indicated; Pulmonary Function Test
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Pulmonary Patients

SUMMARY:
This study was developed in order for the professional-staff at the Pulmonary-Critical Care Medical Branch (PCCMB) of the National Heart, Lung, and Blood Institute to maintain their skills and increase their understanding of lung diseases.

The study will permit PCCMB staff members to evaluate and treat patients with lung disease who do not meet the criteria for other research studies.

DETAILED DESCRIPTION:
The professional staff in the Cardiovascular and Pulmonary Branch (CPB) needs to maintain their clinical skills and to enhance their clinical knowledge. The purpose of this protocol is to permit CPB staff to evaluate and treat patients with pulmonary disease who do not meet the criteria for existing research protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients 8 years old and older with signs or symptoms of pulmonary disease of medical interest to the professional staff of CPB will be eligible for participation in this protocol. Only standard diagnostic procedures and conventional therapy will be performed. Patients will not be subjected to any research procedures. This protocol does not commit the NIH to medical or surgical treatment of protocol participants after discharge. Patients will be discharged to the referring physician.

Consenting to pregnancy testing in minors of childbearing age:

We will inform the minor during the assent process that for safety, we need to do a pregnancy test. She will also be told that if it is positive, we will counsel her and help her tell her parents. If the minor does not want to proceed she will be advised not to sign assent and her enrollment on this training protocol will end.

EXCLUSION CRITERIA:

Patients without symptoms of pulmonary disease will be excluded from this protocol.

Ages: 8 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary disease who do not meet the criteria for existing research protocols.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 1997-02-12 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
to permit PB staff to evaluate and treat patients with pulmonary disease who do not meet the criteria for existing research protocols. | 1 visit
  The purpose of this protocol is to permit PB staff to evaluate and treat patients with pulmonary disease who do not meet the criteria for existing research protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1997-H-0061.html